CLINICAL TRIAL: NCT03930849
Title: Pilot Study of Technology Assisted Depression Treatment Adherence
Brief Title: Pilot Study of Annie Text Messaging for Depression Treatment Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PPO 18-111
Record Dates: First submitted 2019-04-16; First posted 2019-04-29 (Actual); Results first posted 2022-02-18 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Depression
Keywords: Depression; Patient Participation; Text messaging; Patient Portals
MeSH Terms: conditions — Depression; Patient Participation

STUDY DESIGN:
Intervention Model Description: This study will test an intervention designed to improve antidepressant adherence and depression outcomes in Veterans initiating or changing antidepressant medication to treat depression. Veterans will be assigned to 1) use Annie, VA's short message service (SMS) in combination with My HealtheVet, VA's online patient portal, 2) use Annie plus receive a weekly phone call, or 3) to the control group who will not be enrolled in Annie.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- AIMS Intervention (Experimental): Participants randomized to the AIMS arm be enrolled in VA's Annie text messaging program and receive the study protocol.
  Interventions: Behavioral: AIMS
- No Intervention (No Intervention): Participants randomized to the no intervention arm will not be enrolled in the Annie text messaging program.
- AIMS Intervention Plus (Experimental): Participants randomized to the AIMS Intervention Plus arm will be enrolled in VA's Annie text messaging program/study protocol and receive a weekly phone call.
  Interventions: Behavioral: AIMS plus

INTERVENTIONS:
Behavioral: AIMS — Participants randomized to the AIMS arm be enrolled in VA's Annie text messaging program and receive the study protocol. Annie text messages will ask the participate to provide feedback about specific domains related to their depression treatment and goals. The Veteran participant will receive a weekly report about their Annie responses through My HealtheVet, VA's patient portal, and instructed to share information with their care team at their next scheduled appointment. In addition, a summary of response will be provided to the participant's clinician prior to their appointment(s) during the studies 12 week time frame.
  Arms: AIMS Intervention
Behavioral: AIMS plus — Participants randomized to the AIMS Plus arm will receive a weekly phone call in addition to being enrolled in VA's Annie text messaging program/study protocol. Annie text messages will ask the participate to provide feedback about specific domains related to their depression treatment and goals. The Veteran participant will receive a weekly report about their Annie responses through My HealtheVet, VA's patient portal, and instructed to share information with their care team at their next scheduled appointment. In addition, a summary of response will be provided to the participant's clinician prior to their appointment(s) during the studies 12 week time frame.
  Arms: AIMS Intervention Plus

SUMMARY:
Patients and providers need effective tools to help promote adherence to newly prescribed medications for depression and to determine if this medication is improving depressed mood. This study will test an intervention that uses 1) VA's text messaging program called Annie to help patient's engage in self-management when starting a new medication for depression and 2) My HealtheVet, VA's patient portal, for education and communication with their VA health care team. The goals of this intervention are to improve adherence to depression medication and depressive symptoms in Veterans.

DETAILED DESCRIPTION:
Background: There are several known challenges to starting a medication for depression, such as side effects and needing four to six weeks before the effects of the medication may be noticed. This pilot randomized controlled trial will compare usual care to an intervention which aims to improve antidepressant adherence and depression outcomes in Veterans initiating medication to treat depression by using Annie, VA's short messaging services (SMS) application and My HealtheVet, VA's patient portal.

Method: Veterans will be eligible if they are initiating a new antidepressant medication as part of their care at the Iowa City VA primary care or mental health. Veterans will be randomized to one of three groups, usual care or 1 of 2 interventional groups (Annie or Annie plus). Veterans in the intervention groups will 1) receive education about depression and the importance of taking medications as prescribed and 2) receive text messages from "Annie" with information and questions for response. For example, are Veterans taking their medication, is their medication working, and how would they rate their mood. They will also receive weekly reports about their responses to Annie through My HealtheVet, VA's patient portal. In addition, Veterans assigned to Annie Plus will receive a weekly phone call to review progress and to answer any questions. Prior to a participant's scheduled follow-up appointment, a summary of information collected to date via Annie will be made available to the clinical team in the medical record. At the end of the study, participants will be invited to complete a recorded interview about their experiences using the Annie text messaging program and to provide any recommendations for changes. VA providers will also be invited to complete a recorded phone interview about their experience with patients using Annie.

For Veterans randomized to the control condition, research staff will provide education about depression and the importance of taking medications as prescribed. Staff will contact participants in this arm by phone just prior to scheduled follow up visits to discuss any concerns the patient may be experiencing. A sample of Veterans will be asked to complete a recorded interview about their medication management at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

VA Patient

* Diagnosed with depression
* Initiating or changing to a new antidepressant medication
* Cell phone with text messaging capabilities
* Registered with My HealtheVet
* Follow-up appointment with their provider in the next 12 weeks
* Internet access
* English speaking VA Providers: provide care to a study participant

Exclusion Criteria:

* Lack of cell phone access/willingness to receive text messages
* Diagnosis of cognitive disorders, psychotic disorders, bipolar disorder, or active substance abuse.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2019-06-21 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn L Turvey, PhD MS, Principal Investigator — Iowa City VA Health Care System, Iowa City, IA
Locations (1):
- Iowa City VA Health Care System, Iowa City, IA, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No
Original VA funded datasets will be retained on VA servers behind VA firewalls. These data will be provided to interested parties following proper filing and verification of a FOIA request and approval by the Privacy Officer. These data will be maintained as required by VA data retention policies.

REFERENCES:
- [Derived] Turvey C, Fuhrmeister L, Klein D, McCoy K, Moeckli J, Stewart Steffensmeier KR, Suiter N, Van Tiem J. Secure Messaging Intervention in Patients Starting New Antidepressant to Promote Adherence: Pilot Randomized Controlled Trial. JMIR Form Res. 2023 Dec 8;7:e51277. doi: 10.2196/51277. PMID 38064267
- [Derived] Van Tiem J, Moeckli J, Suiter N, Fuhrmeister L, Pham K, Dindo L, Turvey C. "A link to the outside:" Patient perspectives on a mobile texting program to improve depression self-management. Patient Educ Couns. 2021 Sep;104(9):2154-2158. doi: 10.1016/j.pec.2021.02.018. Epub 2021 Feb 11. PMID 33627234

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AIMS Intervention | No Intervention | AIMS Intervention Plus
Started | 17 | 18 | 18
Completed | 13 | 18 | 14
Not Completed | 4 | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AIMS Intervention | No Intervention | AIMS Intervention Plus | Total
Number analyzed (Participants) | 17 | 18 | 18 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.11 (10.65) | 49.55 (14.74) | 47.5 (14.26) | 45.72 (13.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 4 | 15
  Male | 13 | 11 | 14 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 1 | 4
  Not Hispanic or Latino | 15 | 17 | 16 | 48
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 2
  White | 17 | 17 | 17 | 51
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 18 | 18 | 53

OUTCOME MEASURES:

1. Primary Outcome: Medication Adherence at Baseline, 6 Weeks and 12 Weeks
Description: Medication Adherence Rating Scale - 10 item self-report measure of medication taking attitudes, behaviors, and side effects. It is scored on a 0-10 scale with higher scores indicating greater adherence.
Time Frame: Baseline, 6 and 12 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | AIMS Intervention | No Intervention | AIMS Intervention Plus
Number analyzed (Participants) | 13 | 18 | 14
score on a scale
  Baseline | 3.41 (0.46) | 1.32 (0.45) | 2.55 (0.45)
  6-Weeks | 2.66 (0.48) | 1.44 (0.45) | 2.16 (0.47)
  12-Weeks | 2.58 (0.48) | 1.56 (0.45) | 2.57 (0.48)
Statistical Analysis 1: Comparison: AIMS Intervention vs No Intervention; Test type: Other; p = 0.10, Mixed Models Analysis; P-value is for F-value reported below of group x time term in a mixed methods analysis; F-value for Type 3 Fixed, df=4 = 2.01

2. Secondary Outcome: Depressive Symptoms at Baseline, 6 Weeks and 12 Weeks
Description: Patient Health Questionnaire (PHQ-9) - a standard instrument for measuring depressive symptom severity and monitoring treatment outcomes over time. A score of 4 or less indicates minimal depression, 5-9 mild depression, 10-14 moderate depression, 15-19 moderately severe depression, and 20-27 indicates severe depression. The total score may range from 0 -27.
Time Frame: Baseline, 6 and 12 weeks
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | AIMS Intervention | No Intervention | AIMS Intervention Plus
Number analyzed (Participants) | 13 | 18 | 14
units on a scale
  Baseline | 15.41 (1.43) | 13.27 (1.38) | 12.00 (1.38)
  6-Weeks | 13.34 (1.55) | 11.38 (1.38) | 9.29 (1.50)
  12-Weeks | 12.20 (1.58) | 11.45 (1.40) | 8.70 (1.56)
Statistical Analysis 1: Comparison: AIMS Intervention vs No Intervention vs AIMS Intervention Plus; Test type: Superiority; p = 0.90, Mixed Models Analysis; P-value is for F-value reported below of group x time analysis in a mixed methods analysis; F statistic GroupxTime, df=4 = .025

3. Secondary Outcome: Medication Side Effects at Baseline, 6 Weeks, and 12 Weeks
Description: The Frequency, Intensity, and Burden of Side Effects Ratings (FIBSER): The 3-item FIBSER asks about the frequency, severity, and functional impact of antidepressant side effects using a 0 to 6- Likert scale. The prevalence and distribution of scores for each domain will be compared across assessment time points. Higher scores indicate greater side effect burden while lower scores indicate lesser. The range for the total score on the measure can span from 0 to 18. A decline in total score is the desired outcome.
Time Frame: Baseline, 6 and 12 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | AIMS Intervention | No Intervention | AIMS Intervention Plus
Number analyzed (Participants) | 13 | 18 | 14
units on a scale
  Baseline | 6.05 (1.00) | 3.38 (0.97) | 3.55 (0.97)
  6-Weeks | 3.83 (1.11) | 4.88 (0.97) | 1.51 (1.07)
  12-Weeks | 4.06 (1.11) | 3.73 (1.01) | 2.53 (1.14)
Statistical Analysis 1: Comparison: AIMS Intervention vs No Intervention vs AIMS Intervention Plus; Test type: Superiority; p = 0.08, Mixed Models Analysis — P-value of F statistic reported below for mixed methods analysis group*time interaction term; F Value Group x Time, DF=4 = 2.12

ADVERSE EVENTS:
Time Frame: Baseline to 6-months
Arm/Group | AIMS Intervention | No Intervention | AIMS Intervention Plus
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/17 | 0/18 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-30): https://cdn.clinicaltrials.gov/large-docs/49/NCT03930849/Prot_SAP_000.pdf